CLINICAL TRIAL: NCT05849610
Title: An Open Label, Multicenter, Phase 2, Pilot Study, Evaluating Early Treatment With Bispecific T-cell Redirectors (Teclistamab and Talquetamab) in the Frontline Therapy of Newly Diagnosed High-risk Multiple Myeloma
Brief Title: Teclistamab-Daratumumab and Talquestamab-Daratumumab in Newly Diagnosed High-risk Multiple Myeloma
Acronym: GEM-TECTAL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEM-TECTAL
Record Dates: First submitted 2023-02-24; First posted 2023-05-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: High-Risk de Novo Multiple Myeloma
Keywords: High-Risk de novo Multiple Myeloma; Teclistamab; Talquetamab; Daratumumab
MeSH Terms: interventions — daratumumab; Bortezomib; Lenalidomide; talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction VRD-Dara + Intensification Tec-Dara + Maintenance Tec-Dara + ERI Tal-Dara (Experimental): Induction (4 cycles) D-VRD. After Induction, all patients recieve 1st INTENSIFICATION treatment (6 cycles of Tec-Dara). Cycles will be of 28 days (4-week cycles) in duration for daratumumab and for Teclistamab. At the end of 1st Intensification timepoint treatments depends on MRD status:
  1. MRD negative patients in CR at the end of Intensification will receive MAINTENANCE therapy with Tec-Dara continuously for 2 years. Crossover: patients who convert MRD positive or relapse from CR any time during Teclistamab maintenance will receive the same treatment as MRD positive individuals (early rescue intervention, ERI).
  2. MRD positive patients or patients who didn't achieve CR despite MRD negativity, will have ERI (Tal-Dara 6 cycles). MRD and response will be evaluated again after 6 cycles treatment with Tal-Dara. MRD negative patients in CR will receive continuous treatment with Tal-Dara for 2 years.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Teclistamab; Drug: Talquetamab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered by SC injection.
Drug: Bortezomib — Bortezomib dose will be calculated using the patient's actual body surface area (BSA) at baseline and will be administered by subcutaneous (SC) injection.
Drug: Lenalidomide — Lenalidomide will be administered by oral route.
Drug: Teclistamab — Teclistamab will be administered by SC injection.
  Other Names: JNJ-64007957
Drug: Talquetamab — Talquetamab will be administered by subcutaneous (SC) injection.
  Other Names: JNJ-64407564

SUMMARY:
The goal of this Phase 2, open-label, multicenter, non-randomized pilot study is to evaluate the efficacy (in terms of MRD negative CR rate after Intensification therapy) and safety of Tec-Dara (Teclistamab+Daratumumab) and Tal-Dara (Talquetamab+Daratumumab) in de novo high-risk multiple myeloma (DNHRMM) patients.

DETAILED DESCRIPTION:
A total of 30 transplant eligible or elderly fit patients with high risk multiple myeloma will be enrolled

1. Patients will receive a 4-cycle Dara+VRD (daratumumab, bortezomib, lenalidomide, dexamethasone) INDUCTION therapy. Cycles will be of 28 days (4-week cycles) in duration for daratumumab and for VRD.

After the 4-cycle Induction, all patients will receive the 1st INTENSIFICATION treatment which consists of 6 cycles of Tec-Dara. Cycles will be of 28 days (4-week cycles) in duration for daratumumab and for teclistamab.

1st Intsensification, patients will receive a 6-cycle Dara+Teclistamab.

2. At the end of 1st Intensification timepoint treatments depends on MRD status:

2.1) MRD negative patients in CR at the end of Intensification will receive MAINTENANCE therapy with Tec-Dara continuously for 2 years. Cycles will be of 28-days in duration for Tec-Dara. Teclistamab (SC) and daratumumab (SC).

2.2) MRD positive patients or patients who didn't achieve CR despite MRD negativity, will have EARLY RESCUE INTERVENTION (ERI) with Tal-Dara for 6 cycles. MRD and response will be evaluated again after 6 cycles treatment with Tal-Dara. MRD negative patients in CR will receive continuous treatment with Tal-Dara for 2 years.

2.2.1 Early Rescue Intervention with Tal-Dara: Patients who are MRD+ after intensification or who convert from MRD negative into positive or experience a relapse from CR (without fulfilling criteria for disease progression) at any time during Tec-Dara treatment will have ERI with Tal-Dara. Cycles will be of 28 days in duration.

2.2.2. MRD negative patients in CR will receive continuous treatment with Tal-Dara for 2 years. Cycles will be of 28-days of duration for Tal-Dara.

4. SALVAGE therapy: If the patient remains MRD+ or doesn't achieve CR despite MRD negativity after 6 cycles of ERI with Tal-Dara or has disease progression at any time, further treatment will be offered as per the investigation decision outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure nor part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient is ≥ 18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place) at the time of informed consent.
* Patient has documented diagnosis of multiple myeloma according to IMWG diagnostic criteria, with at least one of the following high-risk features:

  1. High-risk FISH: del(17p), t(4;14), t(14;16) and 1q amplifications.
  2. R-ISS 3
  3. Presence of extramedullary disease, defined as presence of paramedullary lesions or extramedullary plasmacytoma.

Note: In order to have a representative population with high-risk features, 50% of patients included will have ultra-high risk disease defined as: i) R-ISS 3; ii) Double hit (at least two high-risk cytogenetic abnormalities); iii) One high-risk cytogenetic abnormality + extramedullary disease.

* Patients eligible for transplant with age ≤ 70 years old (young and transplant-eligible) or patients not eligible for transplant with ECOG-PS modified frailty score of 0-1 (elderly-fit).
* Patient has an ECOG performance status of 0, 1or 2.

Exclusion Criteria:

* Prior or current systemic therapy or SCT for any plasma cell dyscrasia, with the exception of 1 cycle of antimyeloma treatment or the emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment while waiting for results of genetic analysis. A cycle of therapy may include treatment with proteasome inhibitors, immunomodulatory drugs, alkylators and corticosteroids, and/or anti-CD38 monoclonal antibodies (i.e, bortezomib-thalidomide-dexamethasone, D-VTD, bortezomib-lenalidomide-dexamethasone, or bortezomib-cyclophosphamide-dexamethasone, are valid options).
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the NCI-CTCAE Version 5.
* Patient has a diagnosis of primary light chain amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), plasma cell leukemia or active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes) at the time of screening.
* Myelodysplastic syndrome or active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than relapsed/refractory multiple myeloma. The only allowed exceptions are malignancies treated within the last 24 months that are considered completely cured:

  1. Non-muscle invasive bladder cancer (solitary Ta-papillary urothelial neoplasm of low malignancy or low grade, < 3 cm, no carcinoma in situ).
  2. Skin cancer (non-melanoma skin cancers treated with curative therapy or localized melanoma treated with curative surgical resection alone).
  3. Noninvasive cervical cancer.
  4. Localized prostate cancer (M0, N0) with a Gleason score of ≤ 7a, treated locally only (radical prostatectomy/radiation therapy/focal treatment).
  5. Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, localized breast cancer and receiving antihormonal agents.
  6. Other malignancy that is considered cured with minimal risk of recurrence.
* Patient has CNS or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy in terms of Measurable Residual Disease (MRD) negative Complete Remission rate by Next Generation Flow Cytometry after Teclistamab plus Daratumumab intensification. | 22 months approximately
  MRD measured by Next Generation Flow Cytometry (NGF, with a sensitivity level of 10-6) after 6 cycles of Tec-Dara therapy.
Evaluate efficacy in terms of Measurable Residual Disease (MRD) negative Complete Remission rate by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan using the Deauville score, after Tec-Dara intensification. | 22 months approximately
  MRD measured by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan.

SECONDARY OUTCOMES:
To evaluate MRD negative CR rate after Daratumumab plus bortezomib, lenalidomide and dexamethasone (D-VRD) induction. | 16 months approximately
  MRD measured by Next Generation Flow Cytometry.
To evaluate MRD negativity after Teclistamab plus Daratumumab (Tec-Dara) intensification using alternative methods | 22 months approximately
  MRD negative rates measured by Next Generation Sequencing (NGS), and Quantitative Immunoprecipitation Free Light Chain Mass Spectrometry (QIP-FLC-MS) after 6 cycles of Tec-Dara therapy.
To evaluate MRD conversion after early rescue intervention with Talqutamab plus Daratumumab (Tal-Dara) | 4 years approximately
  Percentage of patients converting from positive MRD to negative MRD evaluated by NGF, NGS, QIP-MS-FLC and FDG-PET-CT scan.
To evaluate MRD conversion after Tec-Dara intensification | 22 months approximately
  Percentage of patients converting from positive MRD after D-VRD induction to negative MRD evaluated by NGF, NGS, QIP-MS-FLC and FDGPET-CT scan after Tec-Dara intensification.
To evaluate sustained MRD negativity during maintenance treatment in both Tec-Dara and Tal-Dara treatment arms | 76 months approximately
  Proportion of patients with persistent MRD negative disease at month 6, 12, 18 and 24 of maintenance treatment in both Tec-Dara and TalDara treatment, by NGF, NGS, QIP-MS-FLC and FDG-PET-CT scan and annually thereafter.
To assess reappearance of MRD positivity or relapse from CR in patients during the Tec-Dara treatment. | 46 months
  Proportion of patients relapsing from MRD negative CR to MRD positive or who relapse from CR (not fulfilling criteria for disease progression) during any phase of Tec-Dara treatment (intensification or maintenance).
To assess Time to PFS | 76 months approximately
  PFS is defined as the time from the date of first dose of study drug to the date of first documented disease progression, as defined in the International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first. For subjects who have not progressed and are alive, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy. PFS is measured in months.
To assess Time to EFS | 76 months approximately
  EFS is defined as the time from the date of first dose of study drug to the date of first documentation of an event. Definition of event for EFS calculation is: relapse from CR, conversion from Measurable Residual Disease (MRD) negativity (absence of phenotypically aberrant clonal plasma cells by next generation flow with a sensitivity level of 10-6 using the EuroFlow standard operation procedure and complete metabolic response by PET-CT (Deauville score ≤ 3)) to MRD positivity (presence of phenotypically aberrant clonal plasma cells by next generation flow with a sensitivity level of 10-6 using the EuroFlow standard operation procedure and complete metabolic response by PET-CT (Deauville score ≤ 3)), disease progression or death due to any cause, whichever occurs first. For subjects who have not experience any of these events, data will be censored at the last visit. EFS is measured in months.
To assess Time to TNT | 76 months approximately
  TNT is defined as the time between date of first dose of study drug and the first dose of the next treatment received. TNT is measured in months.
To assess Time to DoR | 76 months approximately
  DoR is the date of initial documentation of a response (Partial Response or better) to the date of first documented evidence of progressive disease, as defined in the International Myeloma Working Group (IMWG) criteria. Relapse from complete response is not considered as disease progression. For subjects who have not progressed, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy. DoR is measured in months
To assess Time to OS | 76 months approximately
  OS is defined as the time from the date of first dose of study drug to the date of the subject's death. If the subject is alive or the vital status is unknown, then the subject's data will be censored at the date the subject was last known to be alive. OS is measured in months.
To assess the safety of the treatment described in the protocol | 76 months approximately
  Incidence of treatment-emergent adverse events
Immune profiling and genetic characterization | 76 months approximately
  Analysis of immune subpopulation and genetic markers

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Lahuerta Palacios, Dr, Study Chair — Hospital Universitario 12 de Octubre; Joan Bladé, Dr, Study Chair — Hospital Clinic of Barcelona; Mª Victoria Mateos, Dr, Study Chair — Hospital Clínico Universitario de Salamanca; Paula Rodríguez Otero, Dr, Study Chair — Clínica Universidad de Navarra; Jesús San Miguel, Dr, Study Chair — Clínica Universidad de Navarra
Locations (10):
- Spain (10):
  - Hospital Germans Trials i Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Doce de Octubre, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - H. Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Santiago (CHUS), Santiago de Compostela
  - Hospital Vírgen del Rocío, Seville
  - Hospital Universitari i Politecnic la Fe, Valencia

REFERENCES:
- [Background] Abecma® (idecabtagene vicleucel) [United States Prescribing Information]. Summit, NJ. Celgene Corporation; 2021.
- [Background] Adams HC 3rd, Stevenaert F, Krejcik J, Van der Borght K, Smets T, Bald J, Abraham Y, Ceulemans H, Chiu C, Vanhoof G, Usmani SZ, Plesner T, Lonial S, Nijhof I, Lokhorst HM, Mutis T, van de Donk NWCJ, Sasser AK, Casneuf T. High-Parameter Mass Cytometry Evaluation of Relapsed/Refractory Multiple Myeloma Patients Treated with Daratumumab Demonstrates Immune Modulation as a Novel Mechanism of Action. Cytometry A. 2019 Mar;95(3):279-289. doi: 10.1002/cyto.a.23693. Epub 2018 Dec 11. PMID 30536810
- [Background] Ariza-Heredia EJ, Chemaly RF. Practical review of immunizations in adult patients with cancer. Hum Vaccin Immunother. 2015;11(11):2606-14. doi: 10.1080/21645515.2015.1062189. Epub 2015 Jun 25. PMID 26110220
- [Background] Atamaniuk J, Gleiss A, Porpaczy E, Kainz B, Grunt TW, Raderer M, Hilgarth B, Drach J, Ludwig H, Gisslinger H, Jaeger U, Gaiger A. Overexpression of G protein-coupled receptor 5D in the bone marrow is associated with poor prognosis in patients with multiple myeloma. Eur J Clin Invest. 2012 Sep;42(9):953-60. doi: 10.1111/j.1365-2362.2012.02679.x. Epub 2012 May 16. PMID 22591013
- [Background] Bai S, Jorga K, Xin Y, Jin D, Zheng Y, Damico-Beyer LA, Gupta M, Tang M, Allison DE, Lu D, Zhang Y, Joshi A, Dresser MJ. A guide to rational dosing of monoclonal antibodies. Clin Pharmacokinet. 2012 Feb 1;51(2):119-35. doi: 10.2165/11596370-000000000-00000. PMID 22257150
- [Background] Bergsagel PL, Mateos MV, Gutierrez NC, Rajkumar SV, San Miguel JF. Improving overall survival and overcoming adverse prognosis in the treatment of cytogenetically high-risk multiple myeloma. Blood. 2013 Feb 7;121(6):884-92. doi: 10.1182/blood-2012-05-432203. Epub 2012 Nov 19. PMID 23165477
- [Background] Brauner-Osborne H, Jensen AA, Sheppard PO, Brodin B, Krogsgaard-Larsen P, O'Hara P. Cloning and characterization of a human orphan family C G-protein coupled receptor GPRC5D. Biochim Biophys Acta. 2001 Apr 16;1518(3):237-48. doi: 10.1016/s0167-4781(01)00197-x. PMID 11311935
- [Background] Burtis CA, Ashwood ER. Tietz textbook of clinical chemistry. 3rd ed. Philadelphia: WB Sauders; 1998.
- [Background] Carpenter RO, Evbuomwan MO, Pittaluga S, Rose JJ, Raffeld M, Yang S, Gress RE, Hakim FT, Kochenderfer JN. B-cell maturation antigen is a promising target for adoptive T-cell therapy of multiple myeloma. Clin Cancer Res. 2013 Apr 15;19(8):2048-60. doi: 10.1158/1078-0432.CCR-12-2422. Epub 2013 Jan 23. PMID 23344265
- [Background] Darce JR, Arendt BK, Chang SK, Jelinek DF. Divergent effects of BAFF on human memory B cell differentiation into Ig-secreting cells. J Immunol. 2007 May 1;178(9):5612-22. doi: 10.4049/jimmunol.178.9.5612. PMID 17442944
- [Background] Delforge M, Ludwig H. How I manage the toxicities of myeloma drugs. Blood. 2017 Apr 27;129(17):2359-2367. doi: 10.1182/blood-2017-01-725705. Epub 2017 Mar 8. PMID 28275090
- [Background] Dimopoulos MA, Moreau P, Terpos E, Mateos MV, Zweegman S, Cook G, Delforge M, Hajek R, Schjesvold F, Cavo M, Goldschmidt H, Facon T, Einsele H, Boccadoro M, San-Miguel J, Sonneveld P, Mey U. Multiple Myeloma: EHA-ESMO Clinical Practice Guidelines for Diagnosis, Treatment and Follow-up. Hemasphere. 2021 Feb 3;5(2):e528. doi: 10.1097/HS9.0000000000000528. eCollection 2021 Feb. No abstract available. PMID 33554050
- [Background] Drayson MT, Bowcock S, Planche T, Iqbal G, Pratt G, Yong K, Wood J, Raynes K, Higgins H, Dawkins B, Meads D, Hulme CT, Monahan I, Karunanithi K, Dignum H, Belsham E, Neilson J, Harrison B, Lokare A, Campbell G, Hamblin M, Hawkey P, Whittaker AC, Low E, Dunn JA; TEAMM Trial Management Group and Trial Investigators. Levofloxacin prophylaxis in patients with newly diagnosed myeloma (TEAMM): a multicentre, double-blind, placebo-controlled, randomised, phase 3 trial. Lancet Oncol. 2019 Dec;20(12):1760-1772. doi: 10.1016/S1470-2045(19)30506-6. Epub 2019 Oct 23. PMID 31668592
- [Background] ECOG-ACRIN Cancer Research Group. ECOG Performance Status Scale. Available at: http://ecogacrin.org/resources/ecog-performance-status. Accessed 28 September 2022.
- [Background] Facon T, Dimopoulos MA, Meuleman N, Belch A, Mohty M, Chen WM, Kim K, Zamagni E, Rodriguez-Otero P, Renwick W, Rose C, Tempescul A, Boyle E, Manier S, Attal M, Moreau P, Macro M, Leleu X, Lorraine Chretien M, Ludwig H, Guo S, Sturniolo M, Tinel A, Silvia Monzini M, Costa B, Houck V, Hulin C, Yves Mary J. A simplified frailty scale predicts outcomes in transplant-ineligible patients with newly diagnosed multiple myeloma treated in the FIRST (MM-020) trial. Leukemia. 2020 Jan;34(1):224-233. doi: 10.1038/s41375-019-0539-0. Epub 2019 Aug 19. PMID 31427722
- [Background] Facon T, Kumar SK, Plesner T, Orlowski RZ, Moreau P, Bahlis N, Basu S, Nahi H, Hulin C, Quach H, Goldschmidt H, O'Dwyer M, Perrot A, Venner CP, Weisel K, Mace JR, Raje N, Tiab M, Macro M, Frenzel L, Leleu X, Ahmadi T, Wang J, Van Rampelbergh R, Uhlar CM, Tromp B, Delioukina M, Vermeulen J, Usmani SZ. Daratumumab, lenalidomide, and dexamethasone versus lenalidomide and dexamethasone alone in newly diagnosed multiple myeloma (MAIA): overall survival results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Nov;22(11):1582-1596. doi: 10.1016/S1470-2045(21)00466-6. Epub 2021 Oct 13. PMID 34655533
- [Background] Faiman B, Bilotti E, Mangan PA, Rogers K; IMF Nurse Leadership Board. Steroid-associated side effects in patients with multiple myeloma: consensus statement of the IMF Nurse Leadership Board. Clin J Oncol Nurs. 2008 Jun;12(3 Suppl):53-63. doi: 10.1188/08.CJON.S1.53-62. PMID 18490257
- [Background] Flockhart DA, Thacker, D., McDonald, C., Desta, Z. The Flockhart Cytochrome P450 Drug-Drug Interaction Table. Division of Clinical Pharmacology, Indiana University School of Medicine (Updated 2021). https://druginteractions.medicine.iu.edu/. Accessed 28 September 2022.
- [Background] Frerichs KA, Broekmans MEC, Marin Soto JA, van Kessel B, Heymans MW, Holthof LC, Verkleij CPM, Boominathan R, Vaidya B, Sendecki J, Axel A, Gaudet F, Pillarisetti K, Zweegman S, Adams HC 3rd, Mutis T, van de Donk NWCJ. Preclinical Activity of JNJ-7957, a Novel BCMAxCD3 Bispecific Antibody for the Treatment of Multiple Myeloma, Is Potentiated by Daratumumab. Clin Cancer Res. 2020 May 1;26(9):2203-2215. doi: 10.1158/1078-0432.CCR-19-2299. Epub 2020 Jan 22. PMID 31969333
- [Background] Frigyesi I, Adolfsson J, Ali M, Christophersen MK, Johnsson E, Turesson I, Gullberg U, Hansson M, Nilsson B. Robust isolation of malignant plasma cells in multiple myeloma. Blood. 2014 Feb 27;123(9):1336-40. doi: 10.1182/blood-2013-09-529800. Epub 2014 Jan 2. PMID 24385542
- [Background] Giri S, Grimshaw A, Bal S, Godby K, Kharel P, Djulbegovic B, Dimopoulos MA, Facon T, Usmani SZ, Mateos MV, Costa LJ. Evaluation of Daratumumab for the Treatment of Multiple Myeloma in Patients With High-risk Cytogenetic Factors: A Systematic Review and Meta-analysis. JAMA Oncol. 2020 Nov 1;6(11):1759-1765. doi: 10.1001/jamaoncol.2020.4338. PMID 32970151
- [Background] Global RPh The Clinician's Ultimate Reference: Corticosteroid - Glucocorticoid Conversion Based on Potency. https://globalrph.com/medcalcs/corticosteroid-converter-based-on-anti-inflammatory-potency/. September 2017. Accessed 16 September 2021
- [Background] Goicoechea I, Puig N, Cedena MT, Burgos L, Cordon L, Vidriales MB, Flores-Montero J, Gutierrez NC, Calasanz MJ, Ramos MM, Lara-Astiaso D, Vilas-Zornoza A, Alignani D, Rodriguez I, Sarvide S, Alameda D, Garces JJ, Rodriguez S, Fresquet V, Celay J, Garcia-Sanz R, Martinez-Lopez J, Oriol A, Rios R, Martin-Sanchez J, Martinez-Martinez R, Sarra J, Hernandez MT, de la Rubia J, Krsnik I, Moraleda JM, Palomera L, Bargay J, Martinez-Climent JA, Orfao A, Rosinol L, Mateos MV, Lahuerta JJ, Blade J, San Miguel J, Paiva B. Deep MRD profiling defines outcome and unveils different modes of treatment resistance in standard- and high-risk myeloma. Blood. 2021 Jan 7;137(1):49-60. doi: 10.1182/blood.2020006731. PMID 32693406
- [Background] Hayden PJ, Roddie C, Bader P, Basak GW, Bonig H, Bonini C, Chabannon C, Ciceri F, Corbacioglu S, Ellard R, Sanchez-Guijo F, Jager U, Hildebrandt M, Hudecek M, Kersten MJ, Kohl U, Kuball J, Mielke S, Mohty M, Murray J, Nagler A, Rees J, Rioufol C, Saccardi R, Snowden JA, Styczynski J, Subklewe M, Thieblemont C, Topp M, Ispizua AU, Chen D, Vrhovac R, Gribben JG, Kroger N, Einsele H, Yakoub-Agha I. Management of adults and children receiving CAR T-cell therapy: 2021 best practice recommendations of the European Society for Blood and Marrow Transplantation (EBMT) and the Joint Accreditation Committee of ISCT and EBMT (JACIE) and the European Haematology Association (EHA). Ann Oncol. 2022 Mar;33(3):259-275. doi: 10.1016/j.annonc.2021.12.003. Epub 2021 Dec 16. PMID 34923107
- [Background] Inoue S, Nambu T, Shimomura T. The RAIG family member, GPRC5D, is associated with hard-keratinized structures. J Invest Dermatol. 2004 Mar;122(3):565-73. doi: 10.1046/j.0022-202X.2004.12628.x. PMID 15086536
- [Background] Karnofsky D, Burchenal J, The clinical evaluation of chemotherapeutic agents in cancer. In: MacLeod C, ed. Evaluation of Chemotherapeutic Agents. New York, NY: Columbia University Press; 1949:191-205.
- [Background] Klinger M, Brandl C, Zugmaier G, Hijazi Y, Bargou RC, Topp MS, Gokbuget N, Neumann S, Goebeler M, Viardot A, Stelljes M, Bruggemann M, Hoelzer D, Degenhard E, Nagorsen D, Baeuerle PA, Wolf A, Kufer P. Immunopharmacologic response of patients with B-lineage acute lymphoblastic leukemia to continuous infusion of T cell-engaging CD19/CD3-bispecific BiTE antibody blinatumomab. Blood. 2012 Jun 28;119(26):6226-33. doi: 10.1182/blood-2012-01-400515. Epub 2012 May 16. PMID 22592608
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Labrijn AF, Meesters JI, de Goeij BE, van den Bremer ET, Neijssen J, van Kampen MD, Strumane K, Verploegen S, Kundu A, Gramer MJ, van Berkel PH, van de Winkel JG, Schuurman J, Parren PW. Efficient generation of stable bispecific IgG1 by controlled Fab-arm exchange. Proc Natl Acad Sci U S A. 2013 Mar 26;110(13):5145-50. doi: 10.1073/pnas.1220145110. Epub 2013 Mar 11. PMID 23479652
- [Background] Lahuerta JJ, Paiva B, Vidriales MB, Cordon L, Cedena MT, Puig N, Martinez-Lopez J, Rosinol L, Gutierrez NC, Martin-Ramos ML, Oriol A, Teruel AI, Echeveste MA, de Paz R, de Arriba F, Hernandez MT, Palomera L, Martinez R, Martin A, Alegre A, De la Rubia J, Orfao A, Mateos MV, Blade J, San-Miguel JF; GEM (Grupo Espanol de Mieloma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Group. Depth of Response in Multiple Myeloma: A Pooled Analysis of Three PETHEMA/GEM Clinical Trials. J Clin Oncol. 2017 Sep 1;35(25):2900-2910. doi: 10.1200/JCO.2016.69.2517. Epub 2017 May 12. PMID 28498784
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245
- [Background] Mateos M-V, Dimopoulos MA, Cavo M, et al. Phase 3 Randomized Study of Daratumumab Plus Bortezomib, Melphalan, and Prednisone (D-VMP) Versus Bortezomib, Melphalan, and Prednisone (VMP) in Newly Diagnosed Multiple Myeloma (NDMM) Patients (Pts) Ineligible for Transplant (ALCYONE). Blood. 2017;130(Suppl 1):LBA-4--LBA-4. http://www.bloodjournal.org/content/130/Suppl_1/LBA-4.
- [Background] Mateos MV, Dimopoulos MA, Cavo M, Suzuki K, Jakubowiak A, Knop S, Doyen C, Lucio P, Nagy Z, Kaplan P, Pour L, Cook M, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Shelekhova T, Yoon SS, Iosava G, Fujisaki T, Garg M, Chiu C, Wang J, Carson R, Crist W, Deraedt W, Nguyen H, Qi M, San-Miguel J; ALCYONE Trial Investigators. Daratumumab plus Bortezomib, Melphalan, and Prednisone for Untreated Myeloma. N Engl J Med. 2018 Feb 8;378(6):518-528. doi: 10.1056/NEJMoa1714678. Epub 2017 Dec 12. PMID 29231133
- [Background] Mateos MV, Nahi H, Legiec W, Grosicki S, Vorobyev V, Spicka I, Hungria V, Korenkova S, Bahlis N, Flogegard M, Blade J, Moreau P, Kaiser M, Iida S, Laubach J, Magen H, Cavo M, Hulin C, White D, De Stefano V, Clemens PL, Masterson T, Lantz K, O'Rourke L, Heuck C, Qin X, Parasrampuria DA, Yuan Z, Xu S, Qi M, Usmani SZ. Subcutaneous versus intravenous daratumumab in patients with relapsed or refractory multiple myeloma (COLUMBA): a multicentre, open-label, non-inferiority, randomised, phase 3 trial. Lancet Haematol. 2020 May;7(5):e370-e380. doi: 10.1016/S2352-3026(20)30070-3. Epub 2020 Mar 23. PMID 32213342
- [Background] Moreau P, Attal M, Hulin C, Arnulf B, Belhadj K, Benboubker L, Bene MC, Broijl A, Caillon H, Caillot D, Corre J, Delforge M, Dejoie T, Doyen C, Facon T, Sonntag C, Fontan J, Garderet L, Jie KS, Karlin L, Kuhnowski F, Lambert J, Leleu X, Lenain P, Macro M, Mathiot C, Orsini-Piocelle F, Perrot A, Stoppa AM, van de Donk NW, Wuilleme S, Zweegman S, Kolb B, Touzeau C, Roussel M, Tiab M, Marolleau JP, Meuleman N, Vekemans MC, Westerman M, Klein SK, Levin MD, Fermand JP, Escoffre-Barbe M, Eveillard JR, Garidi R, Ahmadi T, Zhuang S, Chiu C, Pei L, de Boer C, Smith E, Deraedt W, Kampfenkel T, Schecter J, Vermeulen J, Avet-Loiseau H, Sonneveld P. Bortezomib, thalidomide, and dexamethasone with or without daratumumab before and after autologous stem-cell transplantation for newly diagnosed multiple myeloma (CASSIOPEIA): a randomised, open-label, phase 3 study. Lancet. 2019 Jul 6;394(10192):29-38. doi: 10.1016/S0140-6736(19)31240-1. Epub 2019 Jun 3. PMID 31171419
- [Background] Moreau P, Usmani SZ, Garfall AL, et al. Updated Results from MajesTEC-1: Phase 1/2 Study of Teclistamab, a B-Cell Maturation Antigen x CD3 Bispecific Antibody, in Relapsed/Refractory Multiple Myeloma. Blood. 2021;138(Supplement 1):896. doi:10.1182/blood-2021-147915.
- [Background] Mohyuddin GR, Aziz M, McClune B, Abdallah AO, Qazilbash M. Antibiotic prophylaxis for patients with newly diagnosed multiple myeloma: Systematic review and meta-analysis. Eur J Haematol. 2020 May;104(5):420-426. doi: 10.1111/ejh.13374. Epub 2020 Feb 22. PMID 31880853
- [Background] Munshi NC, Anderson LD Jr, Shah N, Madduri D, Berdeja J, Lonial S, Raje N, Lin Y, Siegel D, Oriol A, Moreau P, Yakoub-Agha I, Delforge M, Cavo M, Einsele H, Goldschmidt H, Weisel K, Rambaldi A, Reece D, Petrocca F, Massaro M, Connarn JN, Kaiser S, Patel P, Huang L, Campbell TB, Hege K, San-Miguel J. Idecabtagene Vicleucel in Relapsed and Refractory Multiple Myeloma. N Engl J Med. 2021 Feb 25;384(8):705-716. doi: 10.1056/NEJMoa2024850. PMID 33626253
- [Background] National Cancer Institute, Division of Cancer Treatment and Diagnosis (US Department of Health and Human Services). Cancer Therapy Evaluation Program: Common Terminology Criteria for Adverse Events. https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm. Last updated 19 April 2021. Accessed 05 October 2022.
- [Background] National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®): Multiple Myeloma, version 4.2022 (14 December 2021). Available at: nccn.org. Accessed 28 December 2021.
- [Background] Novak AJ, Darce JR, Arendt BK, Harder B, Henderson K, Kindsvogel W, Gross JA, Greipp PR, Jelinek DF. Expression of BCMA, TACI, and BAFF-R in multiple myeloma: a mechanism for growth and survival. Blood. 2004 Jan 15;103(2):689-94. doi: 10.1182/blood-2003-06-2043. Epub 2003 Sep 25. PMID 14512299
- [Background] Paiva B, Puig N, Cedena MT, Rosinol L, Cordon L, Vidriales MB, Burgos L, Flores-Montero J, Sanoja-Flores L, Lopez-Anglada L, Maldonado R, de la Cruz J, Gutierrez NC, Calasanz MJ, Martin-Ramos ML, Garcia-Sanz R, Martinez-Lopez J, Oriol A, Blanchard MJ, Rios R, Martin J, Martinez-Martinez R, Sureda A, Hernandez MT, de la Rubia J, Krsnik I, Moraleda JM, Palomera L, Bargay J, Van Dongen JJM, Orfao A, Mateos MV, Blade J, San-Miguel JF, Lahuerta JJ; GEM (Grupo Espanol de Mieloma)/PETHEMA (Programa Para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Group. Measurable Residual Disease by Next-Generation Flow Cytometry in Multiple Myeloma. J Clin Oncol. 2020 Mar 10;38(8):784-792. doi: 10.1200/JCO.19.01231. Epub 2019 Nov 26. PMID 31770060
- [Background] Palumbo A, Rajkumar SV, Dimopoulos MA, Richardson PG, San Miguel J, Barlogie B, Harousseau J, Zonder JA, Cavo M, Zangari M, Attal M, Belch A, Knop S, Joshua D, Sezer O, Ludwig H, Vesole D, Blade J, Kyle R, Westin J, Weber D, Bringhen S, Niesvizky R, Waage A, von Lilienfeld-Toal M, Lonial S, Morgan GJ, Orlowski RZ, Shimizu K, Anderson KC, Boccadoro M, Durie BG, Sonneveld P, Hussein MA; International Myeloma Working Group. Prevention of thalidomide- and lenalidomide-associated thrombosis in myeloma. Leukemia. 2008 Feb;22(2):414-23. doi: 10.1038/sj.leu.2405062. Epub 2007 Dec 20. PMID 18094721
- [Background] Palumbo A, Avet-Loiseau H, Oliva S, Lokhorst HM, Goldschmidt H, Rosinol L, Richardson P, Caltagirone S, Lahuerta JJ, Facon T, Bringhen S, Gay F, Attal M, Passera R, Spencer A, Offidani M, Kumar S, Musto P, Lonial S, Petrucci MT, Orlowski RZ, Zamagni E, Morgan G, Dimopoulos MA, Durie BG, Anderson KC, Sonneveld P, San Miguel J, Cavo M, Rajkumar SV, Moreau P. Revised International Staging System for Multiple Myeloma: A Report From International Myeloma Working Group. J Clin Oncol. 2015 Sep 10;33(26):2863-9. doi: 10.1200/JCO.2015.61.2267. Epub 2015 Aug 3. PMID 26240224
- [Background] Pillarisetti K, Edavettal S, Mendonca M, Li Y, Tornetta M, Babich A, Majewski N, Husovsky M, Reeves D, Walsh E, Chin D, Luistro L, Joseph J, Chu G, Packman K, Shetty S, Elsayed Y, Attar R, Gaudet F. A T-cell-redirecting bispecific G-protein-coupled receptor class 5 member D x CD3 antibody to treat multiple myeloma. Blood. 2020 Apr 9;135(15):1232-1243. doi: 10.1182/blood.2019003342. PMID 32040549
- [Background] San-Miguel J, Usmani SZ, Mateos MV, van de Donk NWCJ, Kaufman JL, Moreau P, Oriol A, Plesner T, Benboubker L, Liu K, Hellemans P, Masterson T, Clemens PL, Luo M, Farnsworth A, Nahi H, Chari A. Subcutaneous daratumumab in patients with relapsed or refractory multiple myeloma: Part 2 of the open-label, multicenter, dose-escalation phase 1b study (PAVO). Haematologica. 2021 Jun 1;106(6):1725-1732. doi: 10.3324/haematol.2019.243790. PMID 32354874
- [Background] Sharma P, Kanapuru B, George B, Lin X, Xu Z, Bryan WW, Pazdur R, Theoret MR. FDA Approval Summary: Idecabtagene Vicleucel for Relapsed or Refractory Multiple Myeloma. Clin Cancer Res. 2022 May 2;28(9):1759-1764. doi: 10.1158/1078-0432.CCR-21-3803. PMID 35046063
- [Background] Smith EL, Harrington K, Staehr M, Masakayan R, Jones J, Long TJ, Ng KY, Ghoddusi M, Purdon TJ, Wang X, Do T, Pham MT, Brown JM, De Larrea CF, Olson E, Peguero E, Wang P, Liu H, Xu Y, Garrett-Thomson SC, Almo SC, Wendel HG, Riviere I, Liu C, Sather B, Brentjens RJ. GPRC5D is a target for the immunotherapy of multiple myeloma with rationally designed CAR T cells. Sci Transl Med. 2019 Mar 27;11(485):eaau7746. doi: 10.1126/scitranslmed.aau7746. PMID 30918115
- [Background] Sonneveld P, Avet-Loiseau H, Lonial S, Usmani S, Siegel D, Anderson KC, Chng WJ, Moreau P, Attal M, Kyle RA, Caers J, Hillengass J, San Miguel J, van de Donk NW, Einsele H, Blade J, Durie BG, Goldschmidt H, Mateos MV, Palumbo A, Orlowski R. Treatment of multiple myeloma with high-risk cytogenetics: a consensus of the International Myeloma Working Group. Blood. 2016 Jun 16;127(24):2955-62. doi: 10.1182/blood-2016-01-631200. Epub 2016 Mar 21. PMID 27002115
- [Background] Tai YT, Anderson KC. Targeting B-cell maturation antigen in multiple myeloma. Immunotherapy. 2015;7(11):1187-99. doi: 10.2217/imt.15.77. Epub 2015 Sep 15. PMID 26370838
- [Background] Usmani SZ, Rodriguez-Otero P, Bhutani M, Mateos MV, Miguel JS. Defining and treating high-risk multiple myeloma. Leukemia. 2015 Nov;29(11):2119-25. doi: 10.1038/leu.2015.209. Epub 2015 Aug 12. PMID 26265183
- [Background] van de Donk NWCJ, Pawlyn C, Yong KL. Multiple myeloma. Lancet. 2021 Jan 30;397(10272):410-427. doi: 10.1016/S0140-6736(21)00135-5. PMID 33516340
- [Background] Voorhees PM, Kaufman JL, Laubach J, Sborov DW, Reeves B, Rodriguez C, Chari A, Silbermann R, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Efebera YA, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Murphy S, Lutska Y, Pei H, Ukropec J, Vermeulen J, de Boer C, Hoehn D, Lin TS, Richardson PG. Daratumumab, lenalidomide, bortezomib, and dexamethasone for transplant-eligible newly diagnosed multiple myeloma: the GRIFFIN trial. Blood. 2020 Aug 20;136(8):936-945. doi: 10.1182/blood.2020005288. PMID 32325490
- [Background] Zamagni E, Nanni C, Dozza L, Carlier T, Bailly C, Tacchetti P, Versari A, Chauvie S, Gallamini A, Gamberi B, Caillot D, Patriarca F, Macro M, Boccadoro M, Garderet L, Barbato S, Fanti S, Perrot A, Gay F, Sonneveld P, Karlin L, Cavo M, Bodet-Milin C, Moreau P, Kraeber-Bodere F. Standardization of 18F-FDG-PET/CT According to Deauville Criteria for Metabolic Complete Response Definition in Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2021 Jan 10;39(2):116-125. doi: 10.1200/JCO.20.00386. Epub 2020 Nov 5. PMID 33151787
- [Background] Zubrod C, et al. Appraisal of methods for the study of chemotherapy in man: Comparative therapeutic trial of nitrogen mustard and thiophosphoramide. Journal of Chronic Diseases; 1960:11:7-33